CLINICAL TRIAL: NCT00040586
Title: Phase II Trial of Monoclonal Antibody J591 in Combination With Low-Dose Interleukin-2 in Patients With Recurrent Prostate Cancer
Brief Title: Phase II Trial of Monoclonal Antibody (J591) in Combination With Low-Dose Subcutaneous Interleukin-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BZL Biologics (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1100-471
Record Dates: First submitted 2002-07-01; First posted 2002-07-02 (Estimated); Last update posted 2007-01-22 (Estimated); Status verified 2002-07

CONDITIONS: Prostatic Neoplasms
Keywords: hormone-refractory
MeSH Terms: conditions — Prostatic Neoplasms | interventions — J591 monoclonal antibody; Interleukin-2

INTERVENTIONS:
Drug: Monoclonal Antibody J591
Drug: Recombinant Interleukin-2

SUMMARY:
The monoclonal antibody J591 is being investigated as therapy for patients with prostate cancer, in combination with recombinant interleukin-2 (Proleukin, Aldesleukin). The study is an open-label, non-randomized phase II study for patients with documented hormone refractory prostate cancer.

DETAILED DESCRIPTION:
In this Phase II, open label study, patients will receive daily low-dose subcutaneous rIL-2 (1.2 x 10^6 IU/m^2/day) continuously beginning on day 1. Patients will receive 3 weeks of IL-2, and on day 22 will receive the monoclonal antibody huJ591 via I.V. (25mg/m^2) for 3 consecutive weeks. Il-2 will be continued for 2 additional weeks for a total of 8 weeks. The 8 week regimen will constitute 1 cycle of therapy. Patients who have responded to therapy or have stable disease will be eligible for additional cycles of therapy.

ELIGIBILITY:
Eligibility Criteria:

* Histologic diagnosis (recent or remote) of prostate adenocarcinoma
* Metastatic or recurrent carcinoma of the prostate defined by abnormal CT or MRI and/or abnormal bone scan and/or rising PSA.
* Rising PSA on 3 serial determinations over a period of > or equal to 2 weeks.
* PSA > or equal to 1.0 at the time of entry.
* If patient is being treated with an LHRH analog the drug: a. must be maintained for the duration of the study or b. must be terminated > or equal to 10 weeks prior to entry (for 28 day depot preparations) or 24 weeks (for 3 month depot preparations).

Exclusion Criteria:

* Prior cytotoxic chemotherapy and/or radiation therapy within 4 weeks of entry.
* History of CNS metastasis, and/or history of seizure and/or stroke.
* Lab values: ANC<1500/mm3; platelet count<100,000/mm3; serum creatinine>2.0; SGOT>2 x normal; bilirubin (total)>1.5; serum calcium> or equal to 11.5.
* Active serious infection not controlled by antibiotics.
* Active angina pectoris or NYHA Class III-IV.
* Karnofsky Performance Status <60.
* Life Expectancy < 3 months.
* Age< 21y.
* Other serious illness(es) involving the cardiac, respiratory, CNS, renal, hepatic or hematological organ systems which might preclude completion of this study or interfere with determination of causality of any adverse effects experienced in this study.
* Untreated thyroid disease, with the exception of treated and stable hyperthyroidism or hypothyroidism for at least 4 weeks prior to entry.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- New York Presbyterian Hospital Medical Oncology/Urology Clinics, New York, New York, United States